CLINICAL TRIAL: NCT03060967
Title: Use of an Innovative and Easy-to-use Tool Based on the Perception of Visual Food Stimuli for Assessing Hedonic and Motivational States in Major Depression.
Brief Title: Assessment of Hedonic and Motivational States in Major Depression ( MOODDIS)
Acronym: MOODDIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: C15-88; C15-88 (Other: Institut National de la Santé Et de la Recherche Médicale)
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Major Depression
Keywords: motivation, instrumental tasks, food-related stimuli, size/time discrimination, major depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depressed patients (Experimental): Computer-based tasks evaluating size and time discrimination capacities of food and control images
  Interventions: Behavioral: Computer-based tasks
- Normal Healthy Volunteers (Experimental): Computer-based tasks evaluating size and time discrimination capacities of food and control images
  Interventions: Behavioral: Computer-based tasks

INTERVENTIONS:
Behavioral: Computer-based tasks — Computer-based tasks designed to assess size and time discrimination capacities of food and control images

SUMMARY:
Major depression is a frequent psychiatric disorder with an estimated lifetime prevalence of 16-17% in the general population. Although its pathophysiology is not completely understood, a large body of literature pleads for a causative role of disturbances in reward processes, referring to: i) the hedonic sensation (i.e. "liking") defined by the pleasure felt after exposure to appetitive stimuli, and ii) the motivation (i.e. "wanting") represented by the ability to initiate and maintain behavioral responses oriented toward appetitive stimuli. the investigators have therefore developed and tested a new experimental computer-based and easy-to-use test intended to provide an objective and quantitative measurement of both hedonic and motivational states in humans. According to the task, the subjects are asked to view and to compare two stimuli, an appetitive one (food pictures) and its devalued counterpart (food pictures in greyscale), at each trial, assessing either the size (task A) or the duration of presentation (task B). From these considerations, the present project aims at using our novel tool to: i) assess the hedonic and motivational state in subjects with major depression, ii) compare their responses with healthy volunteers. The present project should demonstrate that the behavioral tests validated in our laboratory are relevant experimental tools for the diagnostic/clinical assessment and for the phenotypic characterization of depressed patients. The application of the test in the therapeutic context could add further information about the efficacy and relevance of the chosen therapy.

DETAILED DESCRIPTION:
Major depression is a frequent psychiatric disorder with an estimated lifetime prevalence of 16-17% in the general population. Although its pathophysiology is not completely understood, a large body of literature pleads for a causative role of disturbances in reward processes, referring to: i) the hedonic sensation (i.e. "liking") defined by the pleasure felt after exposure to appetitive stimuli, and ii) the motivation (i.e. "wanting") represented by the ability to initiate and maintain behavioral responses oriented toward appetitive stimuli. Several methodological approaches have been used to study hedonic and motivational processes in major depression. Some clinical investigations have tried to explore: i) taste sensitivity, as reflective of hedonic reaction to food stimuli, and ii) time judgment, as indicative of the degree of motivation, which is expected to be low when time is perceived long. However, these studies suffer from serious limitations relied on the frequent utilization of subjective assessment methods. Other authors have instead examined either: i) the processing of emotional information using positive, negative, and neutral faces or words, or ii) the processing of the motivational value of reinforcement, such as monetary cues. These experimental paradigms when coupled with functional neuroimaging allow objectively identifying the anatomo-functional correlates of the internal affective state. However, limited availability and costly procedures characterize the use of functional neuroimaging. the investigators have therefore developed and tested a new experimental computer-based and easy-to-use test intended to provide an objective, implicit and quantitative measurement of both hedonic and motivational states in humans. According to the task, the subjects are asked to view and to compare two stimuli, an appetitive one (food pictures; F) and its devalued counterpart (food pictures in greyscale; D), at each trial, assessing either the size (task A) or the duration of presentation (task B). Geometric figures are used as controls and presented in color (C) or greyscale (D) (1). Both tasks are registered under the French agency for the protection of computer software. Here, the investigators propose to use our novel test to: i) assess the hedonic and motivational state in subjects suffering from major depression ii) compare their responses with healthy volunteers. Responses to the test in depressed patients will be evaluated during two separate experimental sessions under either fasting or satiety conditions.

The present study is expected to begin in February 2017 for a total duration of 36 consecutive months. A sample of 36 patients suffering from major depression will be recruited and compared with 36 healthy normal volunteers. They will be matched on age and sex. During the inclusion visit, information about the study design will be delivered before the written inform consent is collected. Thereafter, the subjects will be screened using the "Association pour la Méthodologie et la Documentation en Psychiatrie" (AMDP) questionnaire, the Mini-International Neuropsychiatric Interview and the Three-Factor Eating Questionnaire for the anamnestic, diagnostic and psychometric (eating behavior) evaluations, respectively. Dietary habits will be recorded with a specific and appropriate instrument used in the National Program Nutrition Health.This will be associated to the assessment of: i) depressive and anxiety symptom.

severity with the Montgomery and Asberg Depression Rating Scale, the Brief Anxiety Scale, and overall functioning with the Global Assessment of Functioning scale in depressed patients; and, ii) neuropsychological functions including cognitive flexibility/psychomotor speed with the Trail making Test (A-B) and visuospatial memory with the Rey-Osterreich Figure Test. To ensure that subjects are familiar with the experimental procedure, the tasks A and B will be explained and the first 5-10 trials will be performed. Two separate experimental sessions will then be conducted, one in satiety and the other after a 6-hour fasting from the breakfast, 3-4 days apart. During each session, the participants will be asked to perform the two validated instrumental tasks in front the screen of a computer. Visual analogue scales (VAS) assessing hunger levels will be completed before each task is performed. A VAS will be also used for the global assessment of appetitive properties of the viewed food images just before the end of the second experimental session. This procedure is adopted to avoid giving to the subject specific information about the exact objectives of the study and therefore to potentially limit biased responses to food images.

ELIGIBILITY:
Inclusion Criteria:

* Depressed patient group

  1. to be between 20- and 60-year-old;
  2. to meet the DSM-5 diagnostic criteria for major depressive disorder;
  3. to experience moderate to severe symptoms interfering with the daily functioning, as indicated by a score above 20 on the Montgomery and Asberg depression scale (MADRS);
  4. to understand and accept the experimental procedure and constraints of the present study;
  5. to give written consent for the participation to the study; and,
  6. to be a beneficiary of or affiliated to a health insurance plan.

Healthy volunteer group

1. to be between 20- and 60-year-old;
2. to be free from any history of psychiatric disorder (substance abuse or alcohol abuse, dependence, mood disorders, etc.) that may require the prescription of long-term psychotropic treatment;
3. to understand and accept the experimental procedure and constraints of the study;

3) to give written consent for the participation to the study; and, 4) to be a beneficiary of or affiliated to a health insurance plan

Exclusion Criteria:

* Depressed patient group

  1. to have a previous history of somatic disease (hypertensive heart disease, Raynaud's syndrome, diabetes, adrenal insufficiency, Cushing's syndrome, peripheral neuropathy, epilepsy ...) or requiring long-term corticosteroid therapy;
  2. to experience serious visual disturbances affecting the visual perception of colors;
  3. to meet the DSM-5 diagnostic criteria for a primary psychiatric disorder such as bipolar disorder, schizophrenia, substance abuse / dependence or alcohol abuse, except for social phobia and generalized anxiety disorder that are commonly comorbid to major depression;
  4. to exhibit a moderate or high suicidal risk, assessed by using the corresponding section of the so-called structured diagnostic psychiatric interview "Mini International Neuropsychiatric Interview" (M.I.N.I. 6.0);
  5. to be exposed to the initiation of an antidepressant treatment with either a selective serotonin reuptake inhibitor or a dual serotonin-norepinephrine reuptake inhibitor within the week prior to the study or to be exposed to a change in the daily dosage of such an ongoing antidepressant treatment within the week preceding the study due to its potential sedative and orexigenic properties;
  6. to be exposed to an antidepressant treatment with antagonists at the presynaptic alpha-2 norepinephrine receptors or with tricyclic agents within the week prior to the study due to their potential sedative and orexigenic properties related to their anti-H1 pharmacological profile;
  7. to be exposed to the initiation of anxiolytic/hypnotic treatment within the week before the study or to be exposed to a change in the daily dosage of such an ongoing anxiolytic/hypnotic treatment within the week prior to the study due to its potential sedative properties in relation with its GABAergic activity;
  8. to be exposed to an antipsychotic treatment within the week prior to the study due to its potential sedative and orexigenic properties related to its anti-H1 pharmacological profile;
  9. to be exposed to alcohol consumption within 2 days before the study
  10. to have a body mass index <18.5 or ≥ 30;
  11. to undergo involuntary hospitalization;
  12. to be a pregnant, parturient or nursing women;
  13. to be a subject deprived of its liberty by judicial or administrative decision
  14. to be a subject under the safeguard measures; and,
  15. to be a subject undergoing an exclusion period for another clinical research

Healthy volunteer group

1. to have a previous history of somatic disorders, including neurological disease;
2. to experience serious visual disturbances affecting the visual perception of colors;
3. to be exposed to alcohol consumption within 2 days before the study
4. to have a body mass index <18.5 or ≥ 25;
5. to undergo involuntary hospitalization;
6. to be a pregnant, parturient or nursing women;
7. to be a subject deprived of its liberty by judicial or administrative decision
8. to be a subject under the safeguard measures; and,
9. to be a subject undergoing an exclusion period for another clinical research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Point of subjective equality (PSE) | From fasting to satiety conditions 3 days apart (days 4 and 7 after inclusion)
  Change in the Point of subjective equality (PSE). The PSE is defined as the ratio "F"/"D" or "C"/"D" for which the stimulus "F" or "C" was judged greater than "D" with a probability of 0.5

SECONDARY OUTCOMES:
Percentage of subjective discrimination (PSD) | From fasting to satiety conditions 3 days apart (days 4 and 7 after inclusion)
  Change in the Percentage of subjective discrimination (PSD). The PSD is defined as the percentage of responses where the stimulus "F" or "C" was judged greater than "D" during the trials where the stimulus "F" or "C" was physically equal to "D", in terms of size or duration of presentation.

CONTACTS AND LOCATIONS:
Locations (1):
- NeuroCentre Magendie INSERM U862, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No